CLINICAL TRIAL: NCT03553914
Title: A Randomized Phase 1-2 Study of PLM60 in Patients With Peripheral T-Cell Lymphoma
Brief Title: PLM60 for Peripheral T Cell Lymphoma (PTCL)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IND Inactive Status
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLM60-MC-1201
Record Dates: First submitted 2018-05-01; First posted 2018-06-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 12 mg/m^2 dose group (Experimental): Subjects will receive PLM60 at 12 mg/m^2 dose.
  Interventions: Drug: PLM60
- 16 mg/m^2 dose group (Experimental): Subjects will receive PLM60 at 16 mg/m^2 dose.
  Interventions: Drug: PLM60
- 20 mg/m^2 dose group (Experimental): Subjects will receive PLM60 at 20 mg/m^2 dose.
  Interventions: Drug: PLM60

INTERVENTIONS:
Drug: PLM60 — PLM60 will be administered via intravenous infusion in 28-day cycles for up to 7 cycles.

SUMMARY:
This is a Phase 1-2, randomized, multicenter, open label study of PLM60 administered via intravenous (IV) infusion in 28 day treatment cycles to adult participants with relapsed or refractory Peripheral T Cell Lymphoma (PTCL).

DETAILED DESCRIPTION:
The study is designed to identify and characterize the safety, tolerability, efficacy, and the PK profile of PLM60 in patients with relapsed or refractory PTCL. Phase 1 will explore multiple dose levels and select a single dose level in Phase 2 to more effectively assess efficacy in the PTCL population.

It is anticipated that up to approximately 30 participants will be enrolled during Phase 1. The actual number enrolled, however, will depend on the number of dose-limiting toxicity (DLT)-evaluable participants that complete the first cycle of therapy. Phase 2 will enroll up to 34 participants at the RP2D, some of whom will have been enrolled during Phase 1.

Consequently, up to approximately 55 participants will be treated in the study as a whole.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent prior to study-related procedures
2. Patients with histologically confirmed relapsed or refractory PTCL, who were treated with at least 2 lines of standard therapy and for whom there is no known effective therapy.
3. Recovered from all toxicity from prior anticancer therapy based on clinical evaluation/ judgement of the Investigator
4. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
5. Participants who have sufficient baseline organ function by laboratory evaluations
6. Left ventricular ejection fraction (LVEF) ≥ 50%
7. Life expectancy ≥ 16 weeks
8. Women of childbearing potential must have a negative pregnancy test prior to study entry, and agree to use adequate contraception from study entry through at least 3 months after the last dose of study drug
9. A male participant must agree to use adequate contraception; or female sexual partner who uses adequate contraception measures from study entry through at least 3 months after the last dose of study drug

Additional Inclusion Criteria for Phase 2:

1. Involved lymph nodes or masses should be measurable in at least 2 perpendicular dimensions and be ≥ 1.5 cm in the longest of the perpendicular dimensions (based on Lugano Classification)
2. Agree to undergo pretreatment bone marrow biopsy and post treatment bone marrow biopsy when required to confirm response

Key Exclusion Criteria:

1. Participants with a history of allergy to anthracyclines or liposomal drugs
2. Prior treatment with mitoxantrone, any anthracycline, or anthacenedione
3. Treatment with doxorubicin (with the exception of pegylated liposomal doxorubicin) with a total cumulative dose > 300 mg/m2, or epirubicin with a total cumulative dose > 500 mg/m2
4. Investigational treatment within 4 weeks of the start of PLM60
5. Prior allogeneic stem cell transplantation
6. Current symptomatic (uncontrolled) central nervous system tumor involvement
7. Certain types of cardiac impairment as defined in the protocol at the time of enrolment
8. Any concurrent active malignancy or concurrent malignancy diagnosis with less than 12 months disease free interval
9. Participants with evidence of an active infection
10. Participants with active bleeding
11. Participants who have had organ transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects experiencing AEs and SAEs after treatment with PLM60 | 8 Months
  Percentage of subjects experiencing AEs and SAEs, by evaluating physical examinations, vital signs, ECOG score, ECGs, ECHO or MUGA scans, and clinical laboratory findings
Overall response rate in patients with PTCL after treatment PLM60 | 19 months
  Assessing the overall response rate (ORR) by Lugano Classification

CONTACTS AND LOCATIONS:
Overall Officials: Study Officials, Study Director — Conjupro Biotherapeutics, Inc.
Locations (2):
- United States (2):
  - Gabrail Cancer Center, Canton, Ohio
  - Gabrial Cancer Center, Canton, Ohio

REFERENCES:
- [Background] Li C, Cui J, Wang C, Li Y, Zhang H, Wang J, Li Y, Zhang L, Zhang L, Guo W, Wang Y. Encapsulation of mitoxantrone into pegylated SUVs enhances its antineoplastic efficacy. Eur J Pharm Biopharm. 2008 Oct;70(2):657-65. doi: 10.1016/j.ejpb.2008.05.019. Epub 2008 Jun 6. PMID 18582570
- [Background] Yang J, Shi Y, Li C, Gui L, Zhao X, Liu P, Han X, Song Y, Li N, Du P, Zhang S. Phase I clinical trial of pegylated liposomal mitoxantrone plm60-s: pharmacokinetics, toxicity and preliminary efficacy. Cancer Chemother Pharmacol. 2014 Sep;74(3):637-46. doi: 10.1007/s00280-014-2523-8. Epub 2014 Jul 18. PMID 25034977